CLINICAL TRIAL: NCT02159898
Title: Prospective, Multicenter, Single Blind, Randomized Study Comparing the EndoMAXX Endoluminal Valve Technology (EVT) Fully Covered Esophageal Stent With Valve to the EndoMAXX Fully Covered Esophageal Stent for Malignant Strictures Requiring Stent Placement Across the Gastroesophageal Junction
Brief Title: EndoMAXX Endoluminal Valve Technology (EVT) Compared to EndoMAXX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merit Medical Systems, Inc. (Industry)
Collaborators: Geisinger Clinic (Other); Medical College of Wisconsin (Other); Indiana University (Other); University of Colorado, Denver (Other); Mayo Clinic (Other); Weill Medical College of Cornell University (Other); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESO-P3-12-02
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Results first posted 2018-06-07 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Malignant Esophageal Strictures
Keywords: Esophageal Cancer; Dysphagia; Regurgitation
MeSH Terms: conditions — Esophageal Neoplasms; Deglutition Disorders; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- EndoMAXX Endoluminal Valve Technology (EVT) (Experimental): EndoMAXX Endoluminal Valve Technology (EVT) Fully Covered Esophageal Stent with Valve
  Interventions: Device: EndoMAXX Endoluminal Valve Technology (EVT)
- EndoMAXX (Active Comparator): EndoMAXX Fully Covered Esophageal Stent
  Interventions: Device: EndoMAXX

INTERVENTIONS:
Device: EndoMAXX Endoluminal Valve Technology (EVT)
  Other Names: EndoMAXX Endoluminal Valve Technology (EVT) Fully Covered Esophageal Stent with Valve
  Arms: EndoMAXX Endoluminal Valve Technology (EVT)
Device: EndoMAXX
  Other Names: EndoMAXX Fully Covered Esophageal Stent
  Arms: EndoMAXX

SUMMARY:
This is a prospective, single blinded, randomized study of EndoMAXX Endoluminal Valve Technology (EVT) Fully Covered Esophageal Stent with Valve for the treatment of malignant strictures of the lower esophagus. The purpose of this study is to evaluate improvement of dysphagia due to esophageal stricture with EndoMAXX Endoluminal Valve Technology (EVT) Fully Covered Esophageal Stent with Valve (investigational device) compared to the EndoMAXX Fully Covered Esophageal Stent (reference device).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age or older
2. Patient (or legal representative) is able to understand and provide signed informed consent
3. Patient has a malignant stricture of the distal esophagus or gastric cardia requiring stent placement across the gastroesophageal junction.

Exclusion Criteria:

1. Patient is unwilling or unable to comply with the follow-up schedule
2. Patient is contraindicated for endoscopic procedure for any reason
3. Patient presents with esophagorespiratory fistula
4. Patient has previously undergone esophageal stenting or esophagectomy
5. Female patient is pregnant, breastfeeding, or premenopausal and not using an effective method of contraception
6. Patient's esophageal tumor length exceeds that which can be treated with a single stent (maximum lesion length 9.5cm)
7. Removal of stent is scheduled to occur within six months
8. Patient has trouble swallowing or experiences regurgitation for reasons which are not related to his/her esophageal cancer
9. Any other factor identified by the Investigator that would disqualify the prospective patient from participation in the study including but not limited to coagulative disorders and anesthetic risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kulwinder DUA, MD, Principal Investigator — Medical College of WI
Locations (7):
- United States (7):
  - University of Colorado Denver, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Indiana University, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Weill Cornell Medical College, New York, New York
  - Geisinger Medical Center, Danville, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Dua KS, DeWitt JM, Kessler WR, Diehl DL, Draganov PV, Wagh MS, Kahaleh M, Wong Kee Song LM, Khara HS, Khan AH, Aburajab MM, Ballard D, Forsmark CE, Edmundowicz SA, Brauer BC, Tyberg A, Buttar NS, Adler DG. A phase III, multicenter, prospective, single-blinded, noninferiority, randomized controlled trial on the performance of a novel esophageal stent with an antireflux valve (with video). Gastrointest Endosc. 2019 Jul;90(1):64-74.e3. doi: 10.1016/j.gie.2019.01.013. Epub 2019 Jan 23. PMID 30684601

RESULTS

PARTICIPANT FLOW:
Groups:
- EndoMAXX EVT: EndoMAXX EVT Fully Covered Esophageal Stent with Valve
  EndoMAXX EVT
- EndoMAXX: EndoMAXX Fully Covered Esophageal Stent
  EndoMAXX
Period: Overall Study
Arm/Group | EndoMAXX EVT | EndoMAXX
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EndoMAXX EVT | EndoMAXX | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 13 | 29
  >=65 years | 14 | 17 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 25 | 27 | 52
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Mellow and Pinkas Dysphagia Score at Baseline and 2 Weeks Following the Treatment
Description: The primary endpoint is to evaluate improvement of dysphagia due to esophageal strictures at 2 weeks following treatment.
  Scale:
  0 = able to eat normal diet / no dysphagia.
  1. = able to swallow some solid foods
  2. = able to swallow only semi solid foods
  3. = able to swallow liquids only
  4. = unable to swallow anything / total dysphagia
Time Frame: 2 Weeks Following Treatment
Population: 1 patient was randomized but not treated and other patients are not included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EndoMAXX EVT | EndoMAXX
Number analyzed (Participants) | 25 | 27
units on a scale | 0.6 (0.7) | 0.6 (0.9)

2. Secondary Outcome: GERD-HRQL
Description: Evaluate symptoms of gastric reflux as assessed by Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) instrument at 4 weeks following treatment.
  Scale:
  0 = No symptom
  1. = Symptoms noticeable but not bothersome
  2. = Symptoms noticeable and bothersome but not every day
  3. = Symptoms bothersome every day
  4. = Symptoms affect daily activity
  5. = Symptoms are incapacitating to do daily activities
Time Frame: 4 Weeks Following Treament
Population: Results at week 4, number of patients analyzed differs from baseline due to inability to continue to follow the patients due to death or lost to follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EndoMAXX EVT: EndoMAXX EVT Fully Covered Esophageal Stent with Valve
Arm/Group | EndoMAXX EVT | EndoMAXX
Number analyzed (Participants) | 17 | 25
units on a scale | 6.4 (5.7) | 6.3 (6.9)

ADVERSE EVENTS:
Time Frame: Adverse Events occurring during the study commencing with the date of treatment through the protocol defined 24 week post-treatment follow-up period, or discontinuation from the study due to study stent removal will be collected.
Arm/Group | EndoMAXX Endoluminal Valve Technology (EVT) | EndoMAXX
All-Cause Mortality (participants affected / at risk) | 12/29 | 10/30
Serious Adverse Events (participants affected / at risk) | 19/29 | 14/30
Other Adverse Events (participants affected / at risk) | 15/29 | 11/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoMAXX Endoluminal Valve Technology (EVT) (N=29) | EndoMAXX (N=30)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 2 (2) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Device Dislocation (General disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Non Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Oesophageal Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) | 1 (1)
Sepsis Syndrome (Infections and infestations) | 1 (1) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Small Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Terminal State (General disorders) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoMAXX Endoluminal Valve Technology (EVT) (N=29) | EndoMAXX (N=30)
Device Dislocation (General disorders) | 14 (14) | 10 (10)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes